CLINICAL TRIAL: NCT03425370
Title: Effect of Replacing Buried Sutures With Tissue Adhesive on Aesthetic Outcome of Surgical Wounds.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Wound dehiscence on tissue adhesive side of 1 wound which developed an infection.
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Michael Kolodney, Dermatology Section Chief, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1710792979
Record Dates: First submitted 2018-01-25; First posted 2018-02-07 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-10

CONDITIONS: Surgical Wound
Keywords: Surgical wounds; Tissue adhesive; Sutures; Wound healing
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Intervention Model Description: Wounds halves will be labeled as A (left/superior) or B (right/inferior), the halves will be randomized to receive either tissue glue or deep sutures. The nurse will refer to the randomization list and inform the surgeon which side of the wound will receive tissue glue and which side will receive deep sutures. Following common practice of wound labeling, side A will always be left or superior from the surgeon's perspective, whereas side B will always be right or inferior from the surgeon's perspective.
  Per randomization, half of the wound will be closed with deep absorbable sutures followed by superficial non-absorbable sutures. The other half of the wound will be closed with superficial non-absorbable sutures followed by tissue glue (Dermabond). Tissue glue will be spread to cover an area extending one cm from the wound margin on both sides.
Who Masked: Outcomes Assessor
Masking Description: The efficacy of intervention methods will be assessed at the 3 month and 6 month follow-ups by having the patient and two blinded observers rate the healing progression of the wound using the POSAS. The observers will be either dermatology faculty or dermatology. The POSAS is a standard metric in measuring wound healing in cutaneous surgery studies since it does not require training but takes into account the scar assessment of the patient and observers. Subsequently, the height and width of the scar will be measured and compared to the surrounding unaffected skin. The assessments of the two blind observers will be averaged.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wound Side A: buried sutures, Wound Side B: tissue adhesive (Experimental): Wounds halves will be labeled as A (left/superior) or B (right/inferior), the halves will be randomized to receive either tissue glue or deep sutures.
  Interventions: Procedure: Closure of surgical wounds using buried sutures or tissue adhesive on aesthetic outcome.
- Wound Side A: tissue adhesive, Wound Side B: buried sutures (Experimental): Wounds halves will be labeled as A (left/superior) or B (right/inferior), the halves will be randomized to receive either tissue glue or deep sutures.
  Interventions: Procedure: Closure of surgical wounds using buried sutures or tissue adhesive on aesthetic outcome.

INTERVENTIONS:
Procedure: Closure of surgical wounds using buried sutures or tissue adhesive on aesthetic outcome. — Effect of replacing buried sutures with tissue adhesive on aesthetic outcome of surgical wounds will be measured using the POSAS.

SUMMARY:
Surgery wounds are typically closed with combination of absorbable stitches placed under the skin and non-absorbable stitched placed at the skin surface. Absorbable sutures can produce unwanted side effects when the body produces a reaction to them. The investigators are conducting a study to determine if absorbable stitches can be replaced but tissue glue applied on the surface of the skin. If participants enroll in the study, the investigators will close one half of the participants wound with absorbable stitches placed under the skin and non-absorbable stitches on the surface. The other half of the wound will be closed with non-absorbable stitches and tissue glue. The appearance of the scar (if any) will then be evaluated at 3- and 6-month follow-ups by two dermatologists (either board-certified dermatologists or dermatology residents) and the patient.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Postoperative defects of at least 3 cm, resulting from either Mohs micrographic surgery or surgical excision
* Willing to give informed consent and return for follow-up visits 3 months and 6 months following surgery

Exclusion Criteria:

* Pregnant
* Unable to understand English
* Mentally impaired
* Incarcerated
* Has nonlinear closures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-01-26 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Rating the healing progression of the wound | 3 months after surgical wound closure
  By observation using the Patient-Observer Scar Assessment Scale (POSAS)
Rating the healing progression of the wound | 6 months after surgical wound closure
  By observation using the Patient-Observer Scar Assessment Scale (POSAS)

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Kolodney, MD, PhD, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University University Town Centre Dermatology Clinic, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-22): https://cdn.clinicaltrials.gov/large-docs/70/NCT03425370/Prot_SAP_000.pdf